CLINICAL TRIAL: NCT04439812
Title: Influence of Positive Margins on Tumour Recurrence and Overall Survival After Gastrectomy for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Pablo Priego, Consultant surgeon MD, PhD. Associate Profesor of Surgery, Hospital Universitario Ramon y Cajal
Other Study IDs: 186/20
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Stomach Neoplasms
Keywords: Gastric cancer; gastrectomy; R1; positive margins; recurrence; overall survival; prognosis
MeSH Terms: conditions — Stomach Neoplasms; Margins of Excision; Recurrence | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- R=0: Patients without positive margins after gastrectomy for gastric cancer
  Interventions: Other: Observation
- R=1: Patients with positive margins after gastrectomy for gastric cancer
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — The primary aim of this study was to evaluate the influence of positive margins on the tumour's recurrence and OS after gastrectomy for GC. The secondary outcome was to analyse the possible confounding factors that could affect the recurrence and OS after gastrectomy.

SUMMARY:
Incidence of positive surgical margins after curative gastrectomy ranges from 1% to 20%. It has been suggested that positive surgical margins is an adverse prognosis factor, with a higher local recurrence and worse overall survival (OS). However, the management of these patients remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients who underwent an oncological gastrectomy due to gastric cancer, between January 2010 and December 2018 at Ramon y Cajal University Hospital.

Exclusion Criteria:

* distant disease (including patients with positive cytology), early postoperative mortality (within 30 days after surgery) and follow-up data not available. Resections in patients with palliative intent were also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all consecutive patients who underwent an oncological gastrectomy due to gastric cancer, between January 2010 and December 2018 at Ramon y Cajal University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
evaluate the influence of positive margins on the tumour's recurrence and OS after gastrectomy for GC | 8 years

SECONDARY OUTCOMES:
The secondary outcome was to analyse the possible confounding factors that could affect the recurrence and OS after gastrectomy. | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Priego, MD, PhD, Principal Investigator — Hospital Universitario Ramón y Cajal

IPD SHARING:
Plan to Share IPD: No